CLINICAL TRIAL: NCT01937013
Title: Impact of Emotional Mimicry and Oxytocin on Frontotemporal Dementia
Acronym: IEMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Elizabeth Finger, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-13-270; 166786 (Other: Health Canada); 103555 (Other: Western HSREB); FTDOXY13EF (Other: Internal)
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Frontotemporal Dementia
Keywords: Frontotemporal Dementia; emotion; oxytocin; fMRI
MeSH Terms: conditions — Frontotemporal Dementia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Oxytocin (Experimental): Participants will be randomized to receive 72 IU intranasal oxytocin on either study visit 2 or 3
  Interventions: Drug: Intranasal oxytocin
- Saline Nasal Mist (Placebo Comparator): Participants will be randomized to receive intranasal saline mist (placebo) on opposite visits from the interventional drug visit 2 or 3
  Interventions: Drug: Saline Nasal Mist

INTERVENTIONS:
Drug: Intranasal oxytocin — Oxytocin can be given intravenously (with a needle) or intranasally (a spray into the nose). The intravenous form of drug is approved by Health Canada for use in pregnancy. The intranasal formulation is not currently approved for use by Health Canada, but is used in Europe to induce labour in pregnant women or aid lactation (breastfeeding). Participants will be randomized to receive 72 IU intranasal oxytocin on either study visit 2 or 3.
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin
Drug: Saline Nasal Mist — Participants will be randomized to receive placebo on either study visit 2 or 3.
  Other Names: Placebo
  Arms: Saline Nasal Mist

SUMMARY:
This study will evaluate the effects on emotions and neural activity of a one time dose of intranasal oxytocin vs. placebo in patients with FTD and healthy controls.

DETAILED DESCRIPTION:
Frontotemporal dementia (FTD) and Pick's disease cause changes in personality, behaviour, and emotional responses. The usual treatments for Frontotemporal dementia focus on reducing agitation and aggressive behaviours. However, these drugs do not help all patients who experience blunting of emotion and loss of empathy. This study will evaluate the effects on emotions and neural activity of a one time dose of intranasal oxytocin vs. placebo in patients with FTD and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Ages 30-85
* meet consensus criteria for probable behavioural variant FTD (bvFTD)

Controls:

* Age and sex matched with patients
* Mini-Mental State Exam (MMSE) scores >27

Exclusion Criteria:

Patients:

* history of stroke
* intracranial haemorrhage or other medical or neurological disorder apart from FTD that could affect cognition
* diagnosis of bipolar disorder or schizophrenia not better accounted for by the diagnosis of FTD
* cognitive impairment that precludes comprehension of task instructions
* contraindication to MRI scanning
* severe language or memory deficits that preclude participation in the study visits and measures
* females who are pregnant or breastfeeding (a pregnancy test will be done on females who have not completed menopause).
* uncontrolled hypertension
* bradycardia (rate <48 bpm) or tachycardia (rate > 100 bpm)
* current use of prostaglandins

Controls:

* history of stroke
* intracranial haemorrhage or other medical or neurological disorder
* diagnosis of bipolar disorder or schizophrenia
* cognitive impairment that precludes comprehension of task instructions
* contraindication to MRI scanning
* severe language or memory deficits that preclude participation in the study visits and measures
* females who are pregnant or breastfeeding (a pregnancy test will be done on females who have not completed menopause).
* uncontrolled hypertension
* bradycardia (rate <48 bpm) or tachycardia (rate > 100 bpm)
* current use of prostaglandins

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) BOLD signal | 2 weeks
  Measures of BOLD (Blood Oxygen-Level Dependent) signal change during oxytocin compared to placebo during functional MRI scans

SECONDARY OUTCOMES:
Cognitive and Emotional Task performance | 2 weeks
  Performance on standardized tasks of emotion processing and cognition

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Finger, M.D., Principal Investigator — LawsonHRI, London Health Sciences Centre, Western University, Schulich School of Medicine; Derek Mitchell, PhD, Principal Investigator — Western University
Locations (1):
- Parkwood Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oliver LD, Stewart C, Coleman K, Kryklywy JH, Bartha R, Mitchell DGV, Finger EC. Neural effects of oxytocin and mimicry in frontotemporal dementia: A randomized crossover study. Neurology. 2020 Nov 10;95(19):e2635-e2647. doi: 10.1212/WNL.0000000000010933. Epub 2020 Sep 22. PMID 32963103